CLINICAL TRIAL: NCT06653959
Title: Safety and Efficacy Study of Precise Transcranial Magnetic Stimulation Based on vlPFC-VTA Individualized Functional Connectivity Localization for the Treatment of Post-stress Sleep Disorders
Brief Title: Precision Transcranial Magnetic Stimulation for Patients With Post-stress Sleep Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20242082
Record Dates: First submitted 2024-10-09; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-04

CONDITIONS: Stress, Psychological; Sleep Initiation and Maintenance Disorders; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active Transcranial Magnetic Stimulation (Active Comparator): The most relevant site of functional connectivity between vlPFC-VTA will be targeted for continuous theta burst stimulation
  Interventions: Device: active Transcranial Magnetic Stimulation
- sham Transcranial Magnetic Stimulation (Placebo Comparator): The most relevant site of functional connectivity between vlPFC-VTA will be targeted for sham continuous theta burst stimulation
  Interventions: Device: sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: active Transcranial Magnetic Stimulation — Based on each individual's MRI data, individualized stimulation targets will be found, and then this will be used for stimulation for 5 consecutive days.
  Arms: active Transcranial Magnetic Stimulation
Device: sham Transcranial Magnetic Stimulation — Based on each individual's MRI data, individualized stimulation targets will be found, and then this will be used for sham stimulation for 5 consecutive days.
  Arms: sham Transcranial Magnetic Stimulation

SUMMARY:
This is a randomized, double-blind controlled study that recruited patients with insomnia problems after suffering a stressful event to undergo individualized transcranial magnetic stimulation

DETAILED DESCRIPTION:
This is a randomized, double-blind controlled study that will recruit patients who have experienced a stressful event and currently exhibit severe sleep problems for transcranial magnetic stimulation. They will be randomly assigned to the trial and control groups and will receive 5 consecutive days of continuous theta-wave stimulation, and before and after the treatment they will be assessed on clinical scales and undergo magnetic resonance examinations as well as sleep monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 60 (both 18 and 60) and of any gender;
2. Experienced a severe traumatic event;
3. Stanford Acute Stress Reaction Questionnaire (SASRQ) ≥40 points;
4. PSQI > 7 points;
5. Good compliance and willingness to undergo this therapy.

Exclusion Criteria:

1. Sleep disorders that can be explained by a primary illness;
2. Concurrent psychotherapy;
3. Those with contraindications to magnetic resonance examination and transcranial magnetic stimulation therapy;
4. Combined with serious cardiovascular, hepatic, renal, digestive, hematopoietic system and other primary diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh sleep quality index (PSQI) scores from baseline to post-treatment | Baseline and treatment day 5
  The Pittsburgh Sleep Quality Index, compiled in 1989 by Dr. Buysse, a psychiatrist at the University of Pittsburgh, and others. It is suitable for patients with sleep disorders to evaluate the quality of their sleep, as well as for the general population to assess the quality of their sleep. The scale consists of 9 questions, of which the first 4 are fill-in-the-blanks and the last 5 are multiple-choice (question 5 contains 10 sub-questions) Change = (treatment day 5 Score -Baseline Score).

SECONDARY OUTCOMES:
Change in Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5 scores from baseline to treatment day 5 | Baseline and treatment day 5
  Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5（PCL-5） is a validated, self-reported instrument assessing PTSD symptom severity over the past week or month period .Possible scores range from 0 to 80 .
  Change = (treatment day 5 Score -Baseline Score).
Change in Stanford Acute Stress Reaction Questionnaire (SASRQ) scores from baseline to treatment day 5 | Baseline and treatment day 5
  The Stanford Acute Stress Reaction Questionnaire (SASRQ) is a commonly used international instrument for assessing acute stress disorders. It consists of 5 dimensions, including alertness, dissociation, avoidance, re-experiencing, and impairment of social functioning, with a total of 30 items, ranging from "not experiencing" to "always experiencing". A total of 30 items, ranging from "no experience" to "always experience", were assigned a score of 0 to 5, with a total score of 0 to 150. The higher the total score, the more severe the acute stress disorder, with a score of ≥40 suggesting a moderate likelihood of acute stress disorder.
  Change = (treatment day 5 Score -Baseline Score).
Change in Hamilton Depression Scale（HAMD-17）scores from baseline to treatment day 5 Score | Baseline and treatment day 5
  Hamilton Depression Scale（HAMD-17） is a commonly used clinical evaluation standard for the severity of depressive symptoms. There are 17 items in total, which can be scored before and after treatment to evaluate the severity of the disease and the treatment effect.Possible scores range from 0 to 52 and the higher the score, the worse the symptom.
  Change = (treatment day 5 Score -Baseline Score).
Change in Hamilton Anxiety Scale scores from baseline to treatment day 5 Score | Baseline and treatment day 5
  Hamilton Anxiety Scale (HAMA）is suitable for assessing the severity of anxiety symptoms. It has 14 items and adopts a 5-level scoring method of 0-4 points.Possible scores range from 0 to 56 and the higher the score, the worse the symptom.
  Change = (treatment day 5 Score -Baseline Score).
Change in Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5 scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  Posttraumatic Stress Disorder Check List for Diagnostic and Statistical Manual of Mental Disorders-5（PCL-5） is a validated, self-reported instrument assessing PTSD symptom severity over the past week or month period .Possible scores range from 0 to 80 .
  Change = (28 days after the end of treatment Score -Baseline Score).
Change in Stanford Acute Stress Reaction Questionnaire (SASRQ) scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  The Stanford Acute Stress Reaction Questionnaire (SASRQ) is a commonly used international instrument for assessing acute stress disorders. It consists of 5 dimensions, including alertness, dissociation, avoidance, re-experiencing, and impairment of social functioning, with a total of 30 items, ranging from "not experiencing" to "always experiencing". A total of 30 items, ranging from "no experience" to "always experience", were assigned a score of 0 to 5, with a total score of 0 to 150. The higher the total score, the more severe the acute stress disorder, with a score of ≥40 suggesting a moderate likelihood of acute stress disorder.
  Change = (28 days after the end of treatment Score -Baseline Score).
Change in Hamilton Depression Scale（HAMD-17）scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  Hamilton Depression Scale（HAMD-17） is a commonly used clinical evaluation standard for the severity of depressive symptoms. There are 17 items in total, which can be scored before and after treatment to evaluate the severity of the disease and the treatment effect.Possible scores range from 0 to 52 and the higher the score, the worse the symptom.
  Change = (28 days after the end of treatment Score -Baseline Score).
Change in Hamilton Anxiety Scale scores from baseline to 28 days after the end of treatment | Baseline and 28 days after the end of treatment
  Hamilton Anxiety Scale (HAMA）is suitable for assessing the severity of anxiety symptoms. It has 14 items and adopts a 5-level scoring method of 0-4 points.Possible scores range from 0 to 56 and the higher the score, the worse the symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Min Cai, PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai M, Zhu Y, Shanley MR, Morel C, Ku SM, Zhang H, Shen Y, Friedman AK, Han MH. HCN channel inhibitor induces ketamine-like rapid and sustained antidepressant effects in chronic social defeat stress model. Neurobiol Stress. 2023 Aug 19;26:100565. doi: 10.1016/j.ynstr.2023.100565. eCollection 2023 Sep. PMID 37664876
- [Background] Luo YJ, Li YD, Wang L, Yang SR, Yuan XS, Wang J, Cherasse Y, Lazarus M, Chen JF, Qu WM, Huang ZL. Nucleus accumbens controls wakefulness by a subpopulation of neurons expressing dopamine D1 receptors. Nat Commun. 2018 Apr 20;9(1):1576. doi: 10.1038/s41467-018-03889-3. PMID 29679009
- [Background] Brunelin J, Jalenques I, Trojak B, Attal J, Szekely D, Gay A, Januel D, Haffen E, Schott-Pethelaz AM, Brault C; STEP Group; Poulet E. The efficacy and safety of low frequency repetitive transcranial magnetic stimulation for treatment-resistant depression: the results from a large multicenter French RCT. Brain Stimul. 2014 Nov-Dec;7(6):855-63. doi: 10.1016/j.brs.2014.07.040. Epub 2014 Aug 7. PMID 25192980
- [Background] Blumberger DM, Maller JJ, Thomson L, Mulsant BH, Rajji TK, Maher M, Brown PE, Downar J, Vila-Rodriguez F, Fitzgerald PB, Daskalakis ZJ. Unilateral and bilateral MRI-targeted repetitive transcranial magnetic stimulation for treatment-resistant depression: a randomized controlled study. J Psychiatry Neurosci. 2016 Jun;41(4):E58-66. doi: 10.1503/jpn.150265. PMID 27269205